CLINICAL TRIAL: NCT04828889
Title: A Prospective Interventional Study to Examine the Effectiveness of Anal Enlargement by Dilators as a Therapeutic Physical Tool in Acute Anal Fissure
Brief Title: Effectiveness of Anal Enlargement by Dilators as a Therapeutic Physical Tool in Acute Anal Fissure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-20-7293-DC-CTIL
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Acute Anal Fissure
Keywords: Anal fissure, anal dilator, anal pain, physiotherapy
MeSH Terms: conditions — Fissure in Ano | interventions — Lateral Internal Sphincterotomy

STUDY DESIGN:
Intervention Model Description: Parallel groups: treatment group( with dilators) versus conservative treatment ( follow up)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- research (Experimental): The subjects in the study group will undergo a series of 4 treatments by 2 certified physiotherapists for pelvic floor treatment that will include instruction in self-use of anal dilators once a week for four weeks. The anal dilation will be performed using Dilatan® anal dilators (Enterprises Sapimed, Alessandria) in varying sizes of 22, 23 and 27 mm. In the first week, a 20 mm dilator will be inserted twice a day for at least 10 minutes. In the second week, a 23 mm extender will be inserted into the anus, twice a day for at least 10 minutes. In the last two weeks, a 27 mm extender will be inserted twice a day for at least 10 minutes. To facilitate the insertion of the extender, patients will use lubricating cream. At the end of each week, patients will meet with a pelvic floor physiotherapist to make sure that the insertion is done properly, that there are no side effects and that it is possible to move on to the next step.
  Interventions: Device: Anal dilators
- waiting (No Intervention): The subjects in the waiting group will be able after a month to choose to undergo surgery or also receive treatment by extenders.
- surgery (Active Comparator): The subjects in the surgery group will undergo surgical treatment only.
  Interventions: Procedure: lateral internal sphincterotomy

INTERVENTIONS:
Device: Anal dilators — Anal sphincter training for relaxation
  Arms: research
Procedure: lateral internal sphincterotomy — lateral internal sphincterotomy is a firmly established method for treating anal fissures.
  Arms: surgery

SUMMARY:
The treatment of anal fissure is mainly surgical. There are complications to this treatment, including damage to the inner anal sphincter and the appearance of fecal incontinence.

Anal dilators are devices that allow gradual enlargement of the anus. To date, the use of these dilators has been in cases of sphincter scarring after a surgical procedure that has caused emptying difficulties. Only recently has the use of anal dilators been tried as a treatment for acute anal fissure.

The study is designated to examine whether healing of the fissure can be achieved by conservative treatment with anal extensions and obviating the need for surgical treatment.

DETAILED DESCRIPTION:
Open prospective study. The study will include 75 patients (men and women) aged 18-85 years who are diagnosed with acute anal fissure and candidates for surgery after conservative treatment failure or recurrence of the problem.

During the waiting period for surgery, which lasted about a month, patients will be divided into three equal-sized groups at random (research, waiting and surgery).

Before the start of treatment and at the end of the waiting and surgery period, all patients will undergo:

1. Anal examination by a proctologist to assess the presence and location of the the fissure
2. Fill out a clinical questionnaire that examines the sensation of pain, burning, itching and bleeding during defecation
3. Fill in the Psychometric properties of a questionnaire (HEMO-FISSQoL) to assess the effect of the fissure on daily functioning
4. Fill out a pain assessment questionnaire (VAS)
5. Fill out a quality of life questionnaire. Only patients with evidence of acute anal fissure in the physical examination will be included in the study.

The subjects in the study group will undergo a series of 4 treatments by 2 certified physiotherapists for pelvic floor treatment that will include instruction in self-use of anal dilators once a week for four weeks. The anal dilation will be performed using 'Dilatan'® anal dilators in varying sizes of 22, 23 and 27 mm. In the first week, a 20 mm dilator will be inserted twice a day for at least 10 minutes. In the second week, a 23 mm dilator will be inserted into the anus, twice a day for at least 10 minutes. In the last two weeks, a 27 mm dilator will be inserted twice a day for at least 10 minutes. To facilitate the insertion of the dilator, patients will use lubricating cream. At the end of each week, patients will meet with a pelvic floor physiotherapist to make sure that the insertion is done properly, that there are no side effects and that it is possible to move on to the next step.

The subjects in the waiting group will be able after a month to choose to undergo surgery or also receive treatment by dilators.

The subjects in the surgery group will undergo surgical treatment only. At the end of the waiting month, a comparison will be made between the indicators of the two groups: research and waiting, in order to evaluate the effectiveness of the treatment in the research group.

In the surgery group, these indices will be examined one month after the surgery

The indices to be examined are:

1. Disappearance of the fissure by proctologist's examination
2. Disappearance of pain, burning, itching and bleeding during defecation
3. Improving the level of pain by using a VAS subjective assessment scale from 1-10
4. Improving the effect of the fissure on daily functioning by using the HEMO-FISSQoL
5. Improving the quality of life of the subjects by using the 36-Item Short Form Survey (SF-36)- Quality of Life Questionnaire Further assessments of the improvement in the quality of life of the subjects in the study group will be made three months and 6 months after the end of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* age 18-85 years
* Must have anal pain during bowel movements
* Must have acute posterior anal fissure
* Must have candidacy for surgery after failure of conservative treatment, or recurrence of the problem.

Exclusion Criteria:

* Concomitant anal pathology (anorectal fistulae,abscesses).
* Previous surgery on the pelvic floor.
* Inflammatory bowel disease
* Inability to sign consent to participate in the study
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Full recovery | 4 weeks
  The incidence of patients who achieved a full recovery of fissure at the end of treatment period

SECONDARY OUTCOMES:
Normal defecation | 4 weeks
  The incidence of patients who achieved normal defecation at the end of the treatment period
Quality of life | 4 weeks
  The incidence of patients who achieved higher score of quality of life at the end of the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Dan Carter, Study Director — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No